CLINICAL TRIAL: NCT04362189
Title: A Randomized, Placebo-Controlled, Double-Blind, Efficacy and Safety Study of Allogeneic HB-adMSCs for the Treatment of COVID-19
Brief Title: Efficacy and Safety Study of Allogeneic HB-adMSCs for the Treatment of COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No need to continue with the availability of the COVID-19 VACCINE
Sponsor: Hope Biosciences Research Foundation (Industry)
Collaborators: River Oaks Hospital and Clinics (Other); United Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBCOV03
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: Coronavirus; Stem cells; Mesenchymal stem cells; Adipose-derived mesenchymal stem cells; MSCs; COVID; SARS-CoV-2; Coronavirus disease
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HB-adMSCs (Experimental): Subjects assigned to this arm will receive 4 intravenous infusions of HB-adMSCs at 100 million cells/dose. HB-adMSC infusions will occur at day 0, 3, 7, and 10.
  Interventions: Biological: HB-adMSC
- Placebo (Placebo Comparator): Subjects assigned to this arm will receive 4 intravenous infusions of placebo (saline solution). Infusions will occur at day 0, 3, 7, and 10.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HB-adMSC — Hope Biosciences allogeneic adipose-derived mesenchymal stem cells
  Arms: HB-adMSCs
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
Hope Biosciences is conducting a research study of an investigational product called allogeneic adipose-derived mesenchymal stem cells (abbreviated as HB-adMSCs) as treatment for patients suspected to have COVID-19. The study purpose is to evaluate the safety and efficacy of four IV infusions of either placebo or HB-adMSCs in subjects with COVID-19.

DETAILED DESCRIPTION:
This is a Phase II, Randomized, Placebo-Controlled, Double-Blinded, Clinical Trial to Assess Efficacy of HB-adMSCs to treat COVID-19 patients. 100 patients will be enrolled. Eligible participants are suspected to have COVID-19 and consent to participate. The primary endpoints of this study are to detect change from baseline in inflammatory markers (IL-6, IL-10, TNF-alpha, C Reactive protein), improving oxygenation, and decreasing time to return to room air (RTRA). In addition, participants will be monitored for overall clinical status by standard clinical laboratories, change from baseline in exploratory markers (D-dimer, myoglobin, troponin, creatinine kinase MB, serum ferritin, CD4:CD8 ratio, CD3-CD56+), time to negative PCR results and clinical improvement according to 7-point ordinal scale, as well as incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Men, and women, over 18 years of age inclusively.
2. Patient is suspected to have COVID-19 infection.
3. Provides consent or consent is given by their legally authorized representative (LAR).
4. Agrees to the collection of venous blood per protocol.
5. Women of childbearing potential (WOCBP) and men (if their sexual partners are WOCBP) must use at least 1 highly effective form of birth control throughout the study and for 6 months after the last dose of study treatment. Highly effective methods of birth control include true sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk, in line with the preferred and usual lifestyle of the patient), surgery (bilateral tubal ligation or occlusion, vasectomized partner), progestogen-only or estrogen/progestogen hormonal contraceptive associated with inhibition of ovulation (oral, patch, injectable, implantable, or intravaginal), intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).

Exclusion Criteria:

1. Pregnancy, lactation and those who are not pregnant but do not take effective contraceptive measures, in women of childbearing age. Absence of pregnancy will be confirmed through urine pregnancy test.
2. Patients who have participated or are participating in a clinical trial of an experimental vaccine for SARS-CoV-2 or coronavirus during the study or within 30 days.
3. Inability to provide informed consent or to comply with study requirements.
4. Patients with the following concomitant or past medical history:

   * Both Hypertension and Diabetes Mellitus.
   * Both Hypertension and Chronic Kidney Disease.
   * Both Diabetes Mellitus and Chronic Kidney Disease.
5. History or evidence of alcohol abuse.
6. History or evidence of consumption of illicit drugs.
7. Patients requiring mechanical ventilation.
8. Patients who are determined by the Principal Investigator to be unsuitable for study enrollment for other reasons.
9. Any medical disease or condition that, in the opinion of the site Principal Investigator or sub-investigator, precludes study participation. Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Thakur, MD, Principal Investigator — River Oaks Hospital and Clinics; Joseph Gathe, MD, Principal Investigator — United Memorial Medical Center
Locations (2):
- United States (2):
  - River Oaks Hospital and Clinics, Houston, Texas
  - United Memorial Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Dios C, Vij R, Kim H, Park H, Chang D. Safety of multiple intravenous infusions of adipose-derived mesenchymal stem cells for hospitalized cases of COVID-19: a randomized controlled trial. Front Med (Lausanne). 2023 Dec 22;10:1321303. doi: 10.3389/fmed.2023.1321303. eCollection 2023. PMID 38188343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 59 subjects were assessed for screening, out of which only 48 were enrolled and 11 failed screening. All 48 were randomized in to the two treatment arms: 100MM HB-adMSCs and placebo. 21 out of 48 randomized subjects discontinued.
Pre-assignment Details: A total of 59 subjects were assessed for screening, out of which only 48 were enrolled and 11 failed screening.
Period: Overall Study
Arm/Group | HB-adMSCs | Placebo
Started | 33 | 15
Completed | 18 | 9
Not Completed | 15 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — FDA Clinical Hold | 7 | 2
Not completed — Discharge or Transfer to other Hospital | 3 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Death | 4 | 1

BASELINE CHARACTERISTICS:
Population: Summary of baseline characteristics for all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | HB-adMSCs | Placebo | Total
Number analyzed (Participants) | 33 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (17.6) | 54.7 (15.8) | 53.7 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 20
  Male | 18 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 22
  Not Hispanic or Latino | 20 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 21 | 11 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: lbs] | 194.6 (48.2) | 194.1 (43.7) | 194.4 (46.3)
Height [Mean (Standard Deviation); unit: in] | 66.5 (3.5) | 66.1 (4.4) | 66.4 (3.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (6.3) | 31.2 (5.9) | 30.9 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Necrosis Factor-Alpha (TNF-alpha)
Description: Change from baseline in Tumor Necrosis Factor-Alpha (TNF-alpha) in the blood (pg/mL)
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
pg/mL
  Day 0 (Baseline) | 15.5 (13.9) | 18.2 (12.3)
  Day 3 | 26.1 (26.5) | 15.9 (10.0)
  Day 7 | 33.4 (49.8) | 35.3 (38.8)
  Day 10 | 20.3 (11.3) | 30.5 (40.5)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = -1.93 — Slope represents beta coefficient for arm * time interaction

2. Primary Outcome: Interleukin-10 (IL-10)
Description: Change from baseline level of Interleukin-10 (IL-10) in the blood (pg/mL)
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
pg/mL
  Day 0 (Baseline) | 16.3 (19.4) | 11.9 (16.6)
  Day 3 | 18.8 (39.1) | 44.7 (98.9)
  Day 7 | 30.8 (86.3) | 27.2 (65.1)
  Day 10 | 13.0 (13.5) | 8.4 (10.8)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Test type: Superiority; Slope = -1.31 — Slope represents beta coefficient for arm * time interaction

3. Primary Outcome: Interleukin-6 (IL-6)
Description: Change from baseline in Interleukin-6 (IL-6) in the blood (pg/mL)
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
pg/mL
  Day 0 (Baseline) | 24.3 (71.8) | 69.4 (166.5)
  Day 3 | 46.3 (104.0) | 376.6 (988.7)
  Day 7 | 65.4 (186.8) | 197.8 (539.7)
  Day 10 | 35.0 (70.4) | 12.4 (23.9)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = 1.36 — Slope represents beta coefficient for arm * time interaction

4. Primary Outcome: C-Reactive Protein (CRP)
Description: Change from baseline in C-Reactive Protein (CRP) in the blood (mg/L)
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mg/L
  Day 0 (Baseline) | 4.9 (5.8) | 3.8 (5.1)
  Day 3 | 4.8 (7.5) | 4.5 (9.2)
  Day 7 | 3.6 (3.4) | 2.2 (4.1)
  Day 10 | 3.5 (4.8) | 0.2 (0.2)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = 0.23 — Slope represents beta coefficient for arm * time interaction

5. Primary Outcome: Oxygenation
Description: Change from baseline Oxygenation (%) in the blood
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: % of Oxygen Saturation
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of Oxygen Saturation
  Day 0 (Baseline) | 95.3 (3.1) | 89.4 (19.1)
  Day 3 | 95.4 (3.2) | 94.5 (4.7)
  Day 7 | 96.2 (2.2) | 95.8 (5.7)
  Day 10 | 96.7 (2.5) | 96.7 (1.7)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = -0.15 — Slope represents beta coefficient for arm * time interaction

6. Primary Outcome: Return To Room Air (RTRA)
Description: Number of participants who returned to room air
Time Frame: Day 0, 3, 7, and 10
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Participants
  Day 0 | 15 | 4
  Day 3 | 13 | 8
  Day 7 | 11 | 7
  Day 10 | 12 | 8
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Odds Ratio (OR) = 0.20 — HB-adMSCs represents Numerator and Placebo represents Denominator

7. Secondary Outcome: D-dimer
Description: Change from baseline in D-dimer in the blood (mg/L)
Time Frame: Day 0, 3, 7, and Day 10
Population: We had 24 participants in the treatment group and 9 in the placebo who had D-dimer values available.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 24 | 9
mg/L
  Day 0 | 1.3 (1.4) | 2.1 (2.6)
  Day 3: number analyzed (Participants) | 16 | 6
  Day 3 | 1.2 (1.7) | 2.3 (2.8)
  Day 7: number analyzed (Participants) | 8 | 2
  Day 7 | 0.7 (0.5) | 13.6 (9.1)
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 6.8 (7.7) |

8. Secondary Outcome: Myoglobin
Description: Clinical lab evaluation of level of Myoglobin in the blood (ng/mL)
Time Frame: Day 0, 3 7, and 10
Population: In the treatment arm, maximum number analyzed was 3 at Day 3 and in Placebo group maximum number analyzed was 1 at Day 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 3 | 1
ng/mL
  Day 0: number analyzed (Participants) | 1 | 1
  Day 0 | 183.0 (NA) — Not enough timepoints analyzed to get a Standard Deviation (SD) value for the HB-adMSCs group. | 21.0 (NA) — Not enough timepoints analyzed to get a Standard Deviation (SD) value for the Placebo group.
  Day 3 | 142.3 (155.8) | 100.0 (NA) — Not enough timepoints analyzed to get a Standard Deviation (SD) value for the Placebo group.
  Day 7: number analyzed (Participants) | 2 | 0
  Day 7 | 21.5 (0.7) |
  Day 10: number analyzed (Participants) | 3 | 0
  Day 10 | 50.3 (48.2) |

9. Secondary Outcome: Troponin
Description: Clinical lab evaluation of level of Troponin in the blood (ng/mL)
Time Frame: Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 14 at Day 0 and in Placebo group maximum number analyzed was 5 at Day 0
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 14 | 5
ng/mL
  Day 0 | 0.5 (1.8) | 0.0 (0.0)
  Day 3: number analyzed (Participants) | 5 | 1
  Day 3 | 0.0 (0.0) | 0.0
  Day 7: number analyzed (Participants) | 7 | 1
  Day 7 | 0.1 (0.2) | 0.0
  Day 10: number analyzed (Participants) | 6 | 0
  Day 10 | 0.0 (0.0) |

10. Secondary Outcome: Creatinine Kinase MB (CK-MB)
Description: Clinical lab evaluation of level of Creatinine Kinase (CK-MB) in the blood (ng/mL)
Time Frame: Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 19 at Day 0 and in Placebo group maximum number analyzed was 8 at Day 0.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 19 | 8
ng/mL
  Day 0 | 2.6 (2.6) | 2.0 (1.1)
  Day 3: number analyzed (Participants) | 9 | 6
  Day 3 | 3.0 (4.6) | 2.2 (1.2)
  Day 7: number analyzed (Participants) | 7 | 2
  Day 7 | 3.3 (2.9) | 2.3 (1.4)
  Day 10: number analyzed (Participants) | 9 | 1
  Day 10 | 3.7 (3.9) | 1.9

11. Secondary Outcome: Serum Ferritin
Description: Clinical lab evaluation of level of Serum Ferritin in the blood (ng/mL)
Time Frame: Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 24 at Day 0 and in Placebo group maximum number analyzed was 7 at Day 0
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 24 | 7
ng/mL
  Day 0 | 420.5 (406.0) | 423.5 (387.9)
  Day 3: number analyzed (Participants) | 12 | 6
  Day 3 | 499.6 (424.2) | 391.2 (324.0)
  Day 7: number analyzed (Participants) | 7 | 2
  Day 7 | 753.9 (449.4) | 361.0 (397.8)
  Day 10: number analyzed (Participants) | 8 | 1
  Day 10 | 509.0 (384.9) | 63.2

12. Secondary Outcome: NK Cell Surface Antigen (CD3-CD56+)
Description: Clinical lab evaluation of Percentage of Cells CD3-CD56+ in the blood (%)
Time Frame: Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 6 at Day 0 and in Placebo group maximum number analyzed was 1 at Day 0
Measure: Mean (Standard Deviation); unit: % of Cells
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 6 | 1
% of Cells
  Day 0 | 66.4 (58.5) | 6.9
  Day 3: number analyzed (Participants) | 0 | 1
  Day 3 |  | 320.0
  Day 7: number analyzed (Participants) | 6 | 0
  Day 7 | 21.9 (30.3) |
  Day 10: number analyzed (Participants) | 0 | 0

13. Secondary Outcome: CD4+/CD8+ Ratio
Description: Clinical lab evaluation of Ratio of CD4+/CD8+ Cells in the blood
Time Frame: Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Ratio
  Day 0 | 2.5 (1.7) | 1.9 (0.9)
  Day 3 | 2.5 (1.3) | 2.6 (1.7)
  Day 7 | 2.4 (1.4) | 2.4 (1.4)
  Day 10 | 2.4 (0.9) | 2.3 (1.3)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = -0.17 — Slope represents beta coefficient for arm * time interaction

14. Secondary Outcome: 7-Point Ordinal Scale
Description: Change from baseline in Ordinal scale score. Scale of 1-7. A score of 1 indicates Death and 7 indicates Subject is not Hospitalized and has no Limitations on activities.
Time Frame: Day 0, 3, 7, 10, and 28 (End of Study)
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Participants
  1: Not hospitalized, no limitations on activities - Day 0 | 1 | 1
  1: Not hospitalized, no limitations on activities - Day 3 | 3 | 3
  1: Not hospitalized, no limitations on activities - Day 7 | 3 | 5
  1: Not hospitalized, no limitations on activities - Day 10 | 6 | 5
  1: Not hospitalized, no limitations on activities - Day 28 (End of Study) | 14 | 7
  2: Not hospitalized, limitation on activities - Day 0 | 2 | 4
  2: Not hospitalized, limitation on activities - Day 3 | 9 | 5
  2: Not hospitalized, limitation on activities - Day 7 | 14 | 7
  2: Not hospitalized, limitation on activities - Day 10 | 12 | 7
  2: Not hospitalized, limitation on activities - Day 28 (End of Study) | 9 | 6
  3: Hospitalized, not requiring supplemental oxygen - Day 0 | 8 | 0
  3: Hospitalized, not requiring supplemental oxygen - Day 3 | 3 | 0
  3: Hospitalized, not requiring supplemental oxygen - Day 7 | 2 | 0
  3: Hospitalized, not requiring supplemental oxygen - Day 10 | 1 | 0
  3: Hospitalized, not requiring supplemental oxygen - Day 28 (End of Study) | 0 | 0
  4: Hospitalized, requiring supplemental oxygen - Day 0 | 15 | 8
  4: Hospitalized, requiring supplemental oxygen - Day 3 | 12 | 6
  4: Hospitalized, requiring supplemental oxygen - Day 7 | 5 | 1
  4: Hospitalized, requiring supplemental oxygen - Day 10 | 4 | 0
  4: Hospitalized, requiring supplemental oxygen - Day 28 (End of Study) | 1 | 0
  5: Hospitalized, on noninvasive ventilation or high flow oxygen devices - Day 0 | 6 | 2
  5: Hospitalized, on noninvasive ventilation or high flow oxygen devices - Day 3 | 4 | 1
  5: Hospitalized, on noninvasive ventilation or high flow oxygen devices - Day 7 | 5 | 1
  5: Hospitalized, on noninvasive ventilation or high flow oxygen devices - Day 10 | 2 | 2
  5: Hospitalized, on noninvasive ventilation or high flow oxygen devices - Day 28 (End of Study) | 0 | 0
  6: Hospitalized, on invasive mechanical ventilation or ECMO - Day 0 | 1 | 0
  6: Hospitalized, on invasive mechanical ventilation or ECMO - Day 3 | 1 | 0
  6: Hospitalized, on invasive mechanical ventilation or ECMO - Day 7 | 0 | 1
  6: Hospitalized, on invasive mechanical ventilation or ECMO - Day 10 | 2 | 0
  6: Hospitalized, on invasive mechanical ventilation or - Day 28 (End of Study) | 1 | 0
  7: Death - Day 0 | 0 | 0
  7: Death - Day 3 | 1 | 0
  7: Death - Day 7 | 4 | 0
  7: Death - Day 10 | 6 | 1
  7: Death - Day 28 (End of Study) | 8 | 2
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = 0.55 — Slope represents beta coefficient for arm * time interaction

15. Secondary Outcome: Computed Tomography (CT) Score
Description: Change from baseline Computed Tomography (CT) Scan Score. A semi-quantitative CT severity scoring was calculated per each of the 5 lobes considering the extent of anatomic involvement: 0, no involvement; 1, < 5% involvement; 2, 5-25% involvement; 3, 26-50% involvement; 4, 51-75% involvement; and 5, > 75% involvement. The resulting global CT score was the sum of each individual lobar score and (0 - no involvement to 25 - maximum involvement). Lower score is better.
Time Frame: Day 0 and Day 28
Measure: Mean (Standard Deviation); unit: Score on a Scale 0-25
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Score on a Scale 0-25
  Day 0 | 2.9 (1.4) | 3.0 (0.9)
  Day 28 | 1.2 (1.6) | 1.2 (1.2)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = 0.26 — Slope represents beta coefficient for arm * time interaction

16. Secondary Outcome: Chest X-Ray Score
Description: Change from baseline in Chest X-Ray Score. Scoring was calculated per each of the 5 lobes considering the extent of anatomic involvement: 0, no involvement; 1, < 5% involvement; 2, 5-25% involvement; 3, 26-50% involvement; 4, 51-75% involvement; and 5, > 75% involvement. The resulting score was the sum of each individual lobar score and (0 - no involvement to 25 - maximum involvement). Lower score is better.
Time Frame: Day 0, Day 28
Measure: Mean (Standard Deviation); unit: Score on a Scale 0-25
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Score on a Scale 0-25
  Day 0 | 2.9 (1.6) | 2.7 (0.6)
  Day 28 | 1.7 (1.6) | 1.5 (2.1)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; Analyses relied on Bayesian inference for test of superiority via generalized linear mixed model; Test type: Superiority; Slope = 0.81 — Slope represents beta coefficient for arm * time interaction

17. Secondary Outcome: Glucose
Description: Clinical lab evaluation of level of Glucose in the blood (mg/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mg/dL
  Screening | 139.3 (58.0) | 148.1 (55.4)
  Day 0 | 153.4 (89.0) | 165.4 (52.5)
  Day 3 | 148.2 (74.8) | 145.6 (58.7)
  Day 7 | 175.7 (106.4) | 165.7 (37.5)
  Day 10 | 166.9 (110.0) | 129.8 (74.4)

18. Secondary Outcome: Blood Urea Nitrogen (BUN)
Description: Clinical lab evaluation of level of Blood Urea Nitrogen (BUN) (mg/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mg/dL
  Screening | 19.7 (14.3) | 14.3 (5.8)
  Day 0 | 22.9 (17.4) | 15.6 (4.8)
  Day 3 | 24.0 (18.5) | 12.7 (4.4)
  Day 7 | 28.4 (28.1) | 19.9 (7.8)
  Day 10 | 19.8 (12.1) | 14.9 (6.0)

19. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) if Non-African American
Description: Clinical lab evaluation of level of Estimated glomerular filtration rate (eGFR) if Non-African American in the blood (mL/min/1.73)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: Estimated glomerular filtration rate (eGFR) if Non-African American
Measure: Mean (Standard Deviation); unit: mL/min/1.73
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 22 | 10
mL/min/1.73
  Screening | 230.3 (270.1) | 127.1 (30.7)
  Day 0: number analyzed (Participants) | 19 | 7
  Day 0 | 143.0 (103.8) | 117.0 (33.9)
  Day 3: number analyzed (Participants) | 14 | 9
  Day 3 | 113.4 (25.2) | 112.8 (22.4)
  Day 7: number analyzed (Participants) | 13 | 6
  Day 7 | 102.8 (44.8) | 109.6 (16.5)
  Day 10: number analyzed (Participants) | 10 | 6
  Day 10 | 107.0 (36.0) | 108.0 (18.0)

20. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) if African American
Description: Clinical lab evaluation of level of Estimated glomerular filtration rate (eGFR) If African American in the blood (mL/min/1.73)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 7 at Day 0 and in Placebo group maximum number analyzed was 2 at Day 10
Measure: Mean (Standard Deviation); unit: mL/min/1.73
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 7 | 2
mL/min/1.73
  Screening: number analyzed (Participants) | 5 | 0
  Screening | 106.4 (37.3) |
  Day 0: number analyzed (Participants) | 7 | 1
  Day 0 | 74.3 (42.7) | 107.0
  Day 3: number analyzed (Participants) | 4 | 1
  Day 3 | 98.2 (58.9) | 97.0
  Day 7: number analyzed (Participants) | 4 | 1
  Day 7 | 78.8 (50.1) | 107.0
  Day 10: number analyzed (Participants) | 5 | 2
  Day 10 | 78.4 (45.7) | 94.5 (26.2)

21. Secondary Outcome: BUN/Creatinine Ratio
Description: Clinical lab evaluation of BUN/Creatinine Ratio in the blood
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Ratio
  Screening | 18.1 (6.6) | 18.9 (2.7)
  Day 0 | 22.9 (11.0) | 20.7 (4.7)
  Day 3 | 22.4 (6.9) | 19.2 (5.8)
  Day 7 | 30.3 (24.6) | 26.1 (8.0)
  Day 10 | 20.2 (7.9) | 18.4 (7.6)

22. Secondary Outcome: Sodium
Description: Clinical lab evaluation of level of Sodium in the blood (mmol/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mmol/L
  Screening | 137.8 (3.5) | 136.9 (3.5)
  Day 0 | 139.4 (3.6) | 137.9 (3.5)
  Day 3 | 140.6 (3.3) | 140.0 (2.8)
  Day 7 | 132.3 (29.6) | 139.3 (3.2)
  Day 10 | 139.2 (4.4) | 141.2 (1.9)

23. Secondary Outcome: Potassium
Description: Clinical lab evaluation of level of Potassium in the blood (mmol/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mmol/L
  Screening | 4.2 (0.5) | 4.2 (0.5)
  Day 0 | 4.1 (0.5) | 4.1 (0.6)
  Day 3 | 3.9 (0.6) | 4.0 (0.3)
  Day 7 | 4.3 (1.3) | 4.5 (0.5)
  Day 10 | 4.5 (1.0) | 4.2 (0.5)

24. Secondary Outcome: Chloride
Description: Clinical lab evaluation of level of Chloride in the blood (mmol/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mmol/L
  Screening | 103.0 (3.9) | 102.2 (2.9)
  Day 0 | 103.3 (3.7) | 101.0 (4.4)
  Day 3 | 103.3 (4.2) | 101.8 (4.1)
  Day 7 | 102.5 (5.5) | 102.1 (2.1)
  Day 10 | 101.9 (4.6) | 104.1 (1.4)

25. Secondary Outcome: Carbon Dioxide Total
Description: Clinical lab evaluation of total level of Carbon Dioxide in the blood (mmol/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mmol/L
  Screening | 25.2 (4.5) | 25.4 (3.1)
  Day 0 | 24.1 (4.8) | 25.3 (4.4)
  Day 3 | 24.6 (4.0) | 25.3 (2.8)
  Day 7 | 23.8 (3.5) | 26.3 (2.8)
  Day 10 | 21.9 (3.8) | 25.4 (3.1)

26. Secondary Outcome: Calcium
Description: Clinical lab evaluation of level of Calcium in the blood (mg/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mg/dL
  Screening | 8.6 (0.5) | 8.7 (0.6)
  Day 0 | 8.4 (0.5) | 8.3 (0.7)
  Day 3 | 8.3 (0.7) | 8.3 (0.8)
  Day 7 | 8.4 (1.1) | 8.7 (0.9)
  Day 10 | 8.6 (1.1) | 9.1 (0.4)

27. Secondary Outcome: Protein Total
Description: Clinical lab evaluation of total level of Protein in the blood (g/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
g/dL
  Screening | 6.2 (0.9) | 6.5 (0.8)
  Day 0 | 5.9 (0.7) | 6.0 (0.8)
  Day 3 | 5.7 (0.8) | 6.0 (0.7)
  Day 7 | 5.6 (1.1) | 6.1 (0.6)
  Day 10 | 6.0 (1.1) | 6.3 (0.4)

28. Secondary Outcome: Albumin
Description: Clinical lab evaluation of level of Albumin in the blood (g/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
g/dL
  Screening | 3.4 (0.5) | 3.6 (0.6)
  Day 0 | 3.4 (0.5) | 3.5 (0.6)
  Day 3 | 3.2 (0.7) | 3.4 (0.6)
  Day 7 | 3.2 (0.8) | 3.5 (0.8)
  Day 10 | 3.4 (0.8) | 3.9 (0.4)

29. Secondary Outcome: Globulin Total
Description: Clinical lab evaluation of the total level of Globulin in the blood (g/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
g/dL
  Screening | 2.8 (0.6) | 2.9 (0.5)
  Day 0 | 2.6 (0.5) | 2.6 (0.4)
  Day 3 | 2.5 (0.5) | 2.6 (0.5)
  Day 7 | 2.5 (0.5) | 2.6 (0.4)
  Day 10 | 2.6 (0.6) | 2.3 (0.4)

30. Secondary Outcome: Albumin/Globulin (A/G) Ratio
Description: Clinical lab evaluation of Albumin/Globulin (A/G) Ratio in the blood
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 14 (at Day 7) and in Placebo group maximum number analyzed was 8 at (Day 10). These were the largest N collected.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 14 | 8
Ratio
  Screening: number analyzed (Participants) | 0 | 0
  Day 0: number analyzed (Participants) | 10 | 4
  Day 0 | 1.4 (0.3) | 1.3 (0.3)
  Day 3: number analyzed (Participants) | 9 | 7
  Day 3 | 1.5 (0.4) | 1.5 (0.4)
  Day 7: number analyzed (Participants) | 14 | 7
  Day 7 | 1.4 (0.3) | 1.4 (0.4)
  Day 10: number analyzed (Participants) | 13 | 8
  Day 10 | 1.3 (0.4) | 1.7 (0.4)

31. Secondary Outcome: Bilirubin Total
Description: Clinical lab evaluation of the total level of Bilirubin in the blood (mg/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
mg/dL
  Screening | 0.6 (0.4) | 0.5 (0.2)
  Day 0 | 0.4 (0.2) | 0.4 (0.3)
  Day 3 | 0.7 (0.8) | 0.4 (0.2)
  Day 7 | 0.5 (0.2) | 0.5 (0.4)
  Day 10 | 0.5 (0.2) | 0.6 (0.5)

32. Secondary Outcome: Alkaline Phosphatase
Description: Clinical lab evaluation of level of Alkaline Phosphatase in the blood (IU/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
IU/L
  Screening | 85.5 (37.2) | 71.9 (19.8)
  Day 0 | 84.9 (35.3) | 66.5 (21.6)
  Day 3 | 101.8 (71.1) | 67.7 (22.1)
  Day 7 | 83.9 (35.0) | 86.6 (15.2)
  Day 10 | 94.2 (47.3) | 79.1 (19.3)

33. Secondary Outcome: Aspartate Aminotransferase (SGOT)
Description: Clinical lab evaluation of level of Aspartate aminotransferase (SGOT) in the blood (IU/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
IU/L
  Screening | 41.9 (33.3) | 41.1 (28.2)
  Day 0 | 30.0 (18.3) | 38.2 (26.4)
  Day 3 | 69.7 (117.3) | 47.3 (33.9)
  Day 7 | 41.4 (52.7) | 46.1 (32.8)
  Day 10 | 36.6 (20.0) | 27.6 (10.1)

34. Secondary Outcome: Alanine Aminotransferase (SGPT)
Description: Clinical lab evaluation of level of Alanine aminotransferase (SGPT) in the blood (IU/L)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
IU/L
  Screening | 50.8 (58.3) | 77.0 (124.5)
  Day 0 | 38.5 (39.7) | 57.2 (38.6)
  Day 3 | 68.0 (78.8) | 107.0 (122.3)
  Day 7 | 46.4 (39.7) | 108.7 (106.2)
  Day 10 | 42.2 (29.3) | 70.8 (83.4)

35. Secondary Outcome: White Blood Count (WBC)
Description: Clinical lab evaluation of count of White Blood Cells (WBCs) in the blood (x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: cells x 10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
cells x 10^3/uL
  Screening | 8.4 (4.0) | 8.6 (5.0)
  Day 0 | 11.3 (10.5) | 10.3 (3.6)
  Day 3 | 13.5 (11.3) | 13.8 (8.7)
  Day 7 | 12.1 (5.8) | 12.7 (5.5)
  Day 10 | 10.4 (5.0) | 11.4 (5.8)

36. Secondary Outcome: Red Blood Cell (RBC) Count
Description: Clinical lab evaluation of Red Blood Cell (RBC) Count in the blood (cells x 10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: cells x 10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
cells x 10^3/uL
  Screening | 4.2 (0.7) | 4.5 (0.6)
  Day 0 | 4.2 (0.8) | 4.5 (1.0)
  Day 3 | 4.1 (0.9) | 4.5 (1.0)
  Day 7 | 3.9 (0.8) | 4.6 (0.8)
  Day 10 | 3.9 (0.9) | 4.3 (0.5)

37. Secondary Outcome: Hemoglobin
Description: Clinical lab evaluation of level of Hemoglobin in the blood (g/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
g/dL
  Screening | 12.0 (2.5) | 12.8 (2.3)
  Day 0 | 11.9 (2.5) | 12.5 (3.1)
  Day 3 | 11.6 (2.7) | 12.1 (2.0)
  Day 7 | 10.8 (2.2) | 13.4 (2.8)
  Day 10 | 11.1 (2.8) | 12.4 (1.7)

38. Secondary Outcome: Hematocrit
Description: Clinical lab evaluation of level of Hematocrit in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: % of RBCs
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of RBCs
  Screening | 37.3 (6.7) | 39.5 (6.3)
  Day 0 | 37.3 (6.8) | 38.8 (8.7)
  Day 3 | 36.0 (7.7) | 38.0 (6.3)
  Day 7 | 33.2 (6.3) | 39.6 (7.8)
  Day 10 | 34.6 (8.3) | 36.7 (4.5)

39. Secondary Outcome: Mean Corpuscular Volume (MCV)
Description: Clinical lab evaluation of level of Mean Corpuscular Volume (MCV) in the blood (fL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
fL
  Screening | 88.8 (9.7) | 86.9 (4.4)
  Day 0 | 89.6 (8.9) | 86.8 (6.0)
  Day 3 | 89.4 (9.8) | 85.8 (6.2)
  Day 7 | 86.8 (9.5) | 85.2 (3.2)
  Day 10 | 89.8 (8.7) | 85.0 (1.9)

40. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH)
Description: Clinical lab evaluation of level of Mean Corpuscular Hemoglobin (MCH) in the blood (pg)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
pg
  Screening | 28.5 (3.9) | 45.4 (67.6)
  Day 0 | 28.6 (3.8) | 27.8 (2.5)
  Day 3 | 28.8 (3.9) | 27.4 (2.9)
  Day 7 | 28.3 (3.9) | 28.7 (1.5)
  Day 10 | 28.7 (3.1) | 28.7 (1.0)

41. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: Clinical lab evaluation of Mean Corpuscular Hemoglobin Concentration (MCHC) in the blood (g/dL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
g/dL
  Screening | 32.0 (1.8) | 32.3 (1.6)
  Day 0 | 31.9 (2.0) | 32.0 (1.8)
  Day 3 | 32.1 (1.9) | 31.8 (1.9)
  Day 7 | 32.6 (2.1) | 33.6 (1.2)
  Day 10 | 31.9 (2.0) | 33.7 (0.8)

42. Secondary Outcome: Red Cell Distribution Width (RDW)
Description: Clinical lab evaluation of Red Cell Distribution Width (RDW) in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: Red Cell Distribution Width %
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Red Cell Distribution Width %
  Screening | 14.4 (1.9) | 13.9 (1.4)
  Day 0 | 18.8 (23.5) | 14.1 (1.5)
  Day 3 | 15.3 (4.8) | 14.3 (2.1)
  Day 7 | 15.5 (4.5) | 13.7 (0.9)
  Day 10 | 14.9 (2.1) | 14.3 (1.2)

43. Secondary Outcome: Platelets
Description: Clinical lab evaluation of level of Platelets in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: cells x 10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
cells x 10^3/uL
  Screening | 232.4 (102.9) | 282.1 (122.8)
  Day 0 | 237.5 (98.8) | 304.8 (101.1)
  Day 3 | 258.2 (115.7) | 295.8 (109.0)
  Day 7 | 273.1 (119.6) | 323.1 (101.2)
  Day 10 | 245.2 (110.5) | 303.8 (86.5)

44. Secondary Outcome: Neutrophils
Description: Clinical lab evaluation of level of Neutrophils in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: % of Neutrophils
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of Neutrophils
  Screening | 78.3 (14.6) | 75.8 (16.1)
  Day 0 | 79.4 (15.4) | 80.7 (11.3)
  Day 3 | 77.0 (15.3) | 75.3 (15.9)
  Day 7 | 73.5 (15.6) | 75.7 (16.6)
  Day 10 | 75.1 (13.3) | 66.2 (17.2)

45. Secondary Outcome: Lymphocytes
Description: Clinical lab evaluation of level of Lymphocytes in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: Percentage of Lymphocytes (%)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Percentage of Lymphocytes (%)
  Screening | 14.4 (11.4) | 16.0 (11.1)
  Day 0 | 11.3 (8.2) | 12.1 (7.9)
  Day 3 | 14.5 (13.9) | 17.2 (12.7)
  Day 7 | 17.4 (13.3) | 16.8 (13.5)
  Day 10 | 17.0 (11.8) | 25.7 (14.2)

46. Secondary Outcome: Monocytes
Description: Clinical lab evaluation of level of Monocytes in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: % of Monocytes
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of Monocytes
  Screening | 5.7 (3.3) | 5.4 (2.7)
  Day 0 | 5.4 (3.6) | 4.9 (2.2)
  Day 3 | 5.4 (2.9) | 5.8 (4.0)
  Day 7 | 5.4 (3.1) | 5.5 (4.8)
  Day 10 | 5.2 (3.6) | 6.5 (3.8)

47. Secondary Outcome: Eosinophils
Description: Clinical lab evaluation of level of Eosinophils n the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: % of Eosinophils
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of Eosinophils
  Screening | 1.1 (3.1) | 0.1 (0.5)
  Day 0 | 0.2 (0.5) | 0.3 (0.5)
  Day 3 | 0.2 (0.6) | 0.8 (1.4)
  Day 7 | 2.5 (9.2) | 0.7 (1.0)
  Day 10 | 1.1 (1.4) | 1.0 (1.1)

48. Secondary Outcome: Basophils
Description: Clinical lab evaluation of level of Basophils in the blood (%)
Time Frame: Screening, Day 0, 3, 7 and 10
Measure: Mean (Standard Deviation); unit: % of Basophils
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
% of Basophils
  Screening | 0.3 (0.4) | 0.1 (0.2)
  Day 0 | 0.1 (0.4) | 0.1 (0.3)
  Day 3 | 0.2 (0.3) | 0.0 (0.0)
  Day 7 | 0.4 (0.7) | 0.8 (0.9)
  Day 10 | 0.4 (0.9) | 0.2 (0.3)

49. Secondary Outcome: Absolute Neutrophils
Description: Clinical lab evaluation of level of Absolute Neutrophils in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at Day screening and in Placebo group maximum number analyzed was 10 at Screening. These were the largest N collected
Measure: Mean (Standard Deviation); unit: cells x 10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 10
cells x 10^3/uL
  Screening | 7.0 (3.8) | 7.5 (4.2)
  Day 0: number analyzed (Participants) | 19 | 6
  Day 0 | 9.7 (10.3) | 7.6 (3.4)
  Day 3: number analyzed (Participants) | 11 | 5
  Day 3 | 15.4 (15.6) | 13.6 (11.5)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 7.4 (4.7) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 5.3 (4.2) |

50. Secondary Outcome: Absolute Lymphocytes
Description: Clinical lab evaluation of level of Absolute Lymphocytes in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 11 at screening. These were the largest N collected for this outcome.
Measure: Mean (Standard Deviation); unit: cells x10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 11
cells x10^3/uL
  Screening | 1.0 (0.6) | 1.1 (1.1)
  Day 0: number analyzed (Participants) | 19 | 6
  Day 0 | 1.0 (0.6) | 1.4 (1.1)
  Day 3: number analyzed (Participants) | 11 | 5
  Day 3 | 1.0 (0.7) | 1.9 (1.4)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 0.8 (0.3) |
  Day 10: number analyzed (Participants) | 5 | 1
  Day 10 | 261.1 (580.8) | 2184.0

51. Secondary Outcome: Absolute Monocytes
Description: Clinical lab evaluation of level of Absolute Monocytes in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 10 at screening.These were the largest N for which data for Absolute Monocytes was collected
Measure: Mean (Standard Deviation); unit: cells x10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 10
cells x10^3/uL
  Screening | 0.4 (0.3) | 0.5 (0.4)
  Day 0: number analyzed (Participants) | 19 | 6
  Day 0 | 1.1 (2.5) | 0.5 (0.4)
  Day 3: number analyzed (Participants) | 11 | 5
  Day 3 | 0.7 (0.5) | 0.8 (0.4)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 0.6 (0.6) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 0.6 (0.4) |

52. Secondary Outcome: Absolute Eosinophils
Description: Clinical lab evaluation of level of Absolute Eosinophils in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 10 at screening.These were the largest N for which data for Absolute Eosinophils was collected
Measure: Mean (Standard Deviation); unit: cells x10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 10
cells x10^3/uL
  Screening | 0.1 (0.3) | 0.0 (0.0)
  Day 0: number analyzed (Participants) | 19 | 6
  Day 0 | 0.0 (0.0) | 0.0 (0.0)
  Day 3: number analyzed (Participants) | 11 | 5
  Day 3 | 0.0 (0.0) | 0.1 (0.2)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 0.0 (0.1) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 0.1 (0.1) |

53. Secondary Outcome: Absolute Basophils
Description: Clinical lab evaluation of level of Absolute Basophils in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 10 at screening.These were the largest N for which data for Absolute Basophils was collected
Measure: Mean (Standard Deviation); unit: cells x10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 10
cells x10^3/uL
  Screening | 0.0 (0.0) | 0.0 (0.0)
  Day 0: number analyzed (Participants) | 19 | 6
  Day 0 | 0.0 (0.0) | 0.0 (0.0)
  Day 3: number analyzed (Participants) | 11 | 5
  Day 3 | 0.0 (0.0) | 0.0 (0.0)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 0.0 (0.0) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 0.0 (0.0) |

54. Secondary Outcome: Immature Granulocytes
Description: Clinical lab evaluation of level of Immature Granulocytes in the blood (%)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 9 at screening. These were the largest N for which data for was collected for Immature granulocytes
Measure: Mean (Standard Deviation); unit: % of Immature Granulocytes
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 9
% of Immature Granulocytes
  Screening | 0.4 (0.6) | 1.2 (1.1)
  Day 0: number analyzed (Participants) | 15 | 5
  Day 0 | 1.0 (1.1) | 1.8 (1.5)
  Day 3: number analyzed (Participants) | 9 | 5
  Day 3 | 1.6 (1.7) | 1.4 (1.1)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 1.0 (0.8) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 0.6 (0.5) |

55. Secondary Outcome: Absolute Immature Granulocytes
Description: Clinical lab evaluation of level of Absolute Immature Granulocytes in the blood (cells x10^3/uL)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 21 at screening and in Placebo group maximum number analyzed was 9 at screening.These were the largest N for which data was collected for Absolute Immature Granulocytes
Measure: Mean (Standard Deviation); unit: cells x10^3/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 21 | 9
cells x10^3/uL
  Screening | 0.0 (0.0) | 0.1 (0.2)
  Day 0: number analyzed (Participants) | 15 | 5
  Day 0 | 0.1 (0.2) | 0.2 (0.2)
  Day 3: number analyzed (Participants) | 9 | 5
  Day 3 | 0.2 (0.2) | 0.3 (0.5)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 0.1 (0.0) |
  Day 10: number analyzed (Participants) | 5 | 0
  Day 10 | 0.0 (0.1) |

56. Secondary Outcome: International Normalized Ratio (INR)
Description: Clinical lab evaluation of International Normalized Ratio (INR)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
Ratio
  Screening | 1.1 (0.1) | 1.1 (0.1)
  Day 0 | 1.2 (0.3) | 1.1 (0.1)
  Day 3 | 1.2 (0.3) | 1.1 (0.1)
  Day 7 | 1.2 (0.4) | 1.1 (0.1)
  Day 10 | 1.4 (0.6) | 1.1 (0.2)

57. Secondary Outcome: Prothrombin Time (PT)
Description: Clinical lab evaluation of Prothrombin Time (seconds)
Time Frame: Screening, Day 0, 3, 7, and 10
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 33 | 15
seconds
  Screening | 11.5 (1.2) | 12.0 (1.4)
  Day 0 | 14.3 (3.9) | 12.9 (2.0)
  Day 3 | 14.4 (3.1) | 13.9 (2.0)
  Day 7 | 15.3 (4.1) | 14.6 (1.4)
  Day 10 | 16.1 (5.8) | 14.3 (1.7)

58. Secondary Outcome: Partial Thromboplastin Time (PTT)
Description: Clinical lab evaluation of Partial Thromboplastin Time (PTT) (seconds)
Time Frame: Screening, Day 0, 3, 7, and 10
Population: In the treatment arm, maximum number analyzed was 25 at screening and in Placebo group maximum number analyzed was11 at screening. These were the largest N for which data for was collected for Partial Thromboplastin time
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 25 | 11
seconds
  Screening | 32.0 (5.5) | 30.4 (3.8)
  Day 0: number analyzed (Participants) | 12 | 6
  Day 0 | 31.6 (6.6) | 29.8 (4.2)
  Day 3: number analyzed (Participants) | 12 | 2
  Day 3 | 32.2 (5.8) | 26.5 (6.4)
  Day 7: number analyzed (Participants) | 4 | 0
  Day 7 | 31.0 (6.9) |
  Day 10: number analyzed (Participants) | 6 | 2
  Day 10 | 24.5 (12.7) | 28.2 (1.4)

ADVERSE EVENTS:
Time Frame: Screening through Day 28 (End of Study)
Description: Out of 48 total subjects, 39 subjects had reported at least one adverse event (AE). A total of 119 AEs were recorded during the entire course of study, out of which 105 were mild in severity, 2 moderate, 1 severe, 1 life threatening, and 10 fatal (death). There were 12 serious adverse events (SAEs) reported during the study period.
Arm/Group | HB-adMSCs | Placebo
All-Cause Mortality (participants affected / at risk) | 8/33 | 2/15
Serious Adverse Events (participants affected / at risk) | 9/33 | 2/15
Other Adverse Events (participants affected / at risk) | 27/33 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=33) | Placebo (N=15)
Cardiopulmonary Failure (Cardiac disorders) | 6 (6) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=33) | Placebo (N=15)
Body Aches (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 3 (4)
Hyperthermia (Nervous system disorders) | 4 (6) | 2 (2)
Fatigue (Nervous system disorders) | 2 (2) | 4 (4)
Anxiety (Nervous system disorders) | 4 (4) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Chest Discomfort (Cardiac disorders) | 1 (1) | 2 (2)
Chills (Nervous system disorders) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vesicular Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Nervous system disorders) | 0 (0) | 1 (1)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Endocrine disorders) | 0 (0) | 1 (1)
Poor Venous Access (Vascular disorders) | 1 (1) | 1 (1)
ESR Raised (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myofascial Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain Natriuretic Peptide Increased (Nervous system disorders) | 1 (1) | 0 (0)
Carbon Dioxide Abnormal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urine Abnormality (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocardial Necrosis Marker Increased (Cardiac disorders) | 1 (1) | 0 (0)
Abnormal Blood Electrolytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Elevated WBC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusional State (Nervous system disorders) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling Abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Kidney Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Puncture Site Bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04362189/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04362189/SAP_001.pdf